CLINICAL TRIAL: NCT04304781
Title: Phase 1 In-vivo Study of KSP/QRH Heptapeptide Dimer for Detection of Biliary Intra-epithelial Neoplasia
Brief Title: Phase 1 In-vivo Biliary Study of KSP/QRH Heptapeptide Dimer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to lack of dimer.
Sponsor: Danielle Kim Turgeon (Other)
Responsible Party: Sponsor-Investigator, Danielle Kim Turgeon, Professor of Internal Medicine and Clinical Track Faculty Ombuds, Medical School, Int Med-Gastroenterology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HUM00173620
Record Dates: First submitted 2020-02-19; First posted 2020-03-11 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dimer Application with SFE imaging (Experimental): Subjects having a standard-of-care ERCP will have the dimer sprayed on an area of interest in the bile duct and images taken with the SFE.
  Interventions: Drug: KSP/QRH dimer

INTERVENTIONS:
Drug: KSP/QRH dimer — Peptide 919288G, Lot No. 17081402, Molecular Weight 3577.0, ≥95% purity. Stored at <20°C. Dark green, lyophilized powder in single-use amber vials.

SUMMARY:
The overall aim of this feasibility study is to develop new technologies for improved detection of cholangiocarcinoma using the SFE-based molecular-imaging mini-cholangioscope (MC) system. This study will combine the use of a fluorescent-labeled peptide dimer that binds specifically to know biomarkers of cholangiocarcinoma for use as a novel imaging agent to guide endoscopic biopsies. This Phase 1B study will be used to provide early evidence of efficacy for the topical application of a peptide dimer that binds to molecular targets that are specific for biliary intra-epithelial neoplasia. A dimer is needed because cancer in the biliary tract is genetically heterogeneous. QRH binds specifically to Epidermal Growth Factor Receptor (EGFR), and KSP binds specifically to Human Epithelial Growth Factor Receptor (HER2). The study will look at peptide binding in subjects having a medical condition requiring an ERCP to diagnose a potential biliary disorder. The Phase 1A first-in-human studies of safety with topical administration by ingestion of KSP/QRH dimer (HUM00141420) has been completed.

ELIGIBILITY:
Inclusion Criteria:

Subject meets all of the following criteria:

* Scheduled for an outpatient ERCP to diagnose a potential biliary disorder (such as an indeterminate biliary stricture)
* Subject is medically cleared for the procedure (e.g. washout for anticoagulants, co-morbidities)
* Age 18 to 100 years
* Willing and able to sign informed consent

Exclusion Criteria:

* Subjects with known allergy or negative reaction to any components of the study drug (list these)
* Subjects on active chemotherapy or radiation treatment
* Pregnant or trying to conceive
* Anything that, in the opinion of the investigator, would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Contrast in Cell Fluorescence | During and immediately after procedure, generally no more than 2 hours
  The fluorescence intensity will be measured by the target/background (T/B) ratio from suspicious regions of bile duct where the fluorescent-labeled peptide is administered. The intensity of the fluorescence of the abnormal tissue compared to the background tissue intensity will be analyzed using statistical analysis for significance comparing the tissue groups' mean T/B ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kim Turgeon, MD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No